CLINICAL TRIAL: NCT06186076
Title: An Open Label, Multicenter, Phase 1/2 Study to Explore the Safety, Tolerability, Pharmacokinetics, and Anti-tumor Activity of TRX-221 in the Treatment of Patients With EGFR Mutant NSCLC Who Progressed Following Prior Therapy With EGFR TKI
Brief Title: A Study to Investigate Safety, Tolerability, PK and Anti-tumor Activity of TRX-221 in EGFRm NSCLC Patients
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Therapex Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TRX-221-001
Record Dates: First submitted 2023-12-06; First posted 2023-12-29 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Carcinoma, Non-Small-Cell Lung; EGFR Mutant Advanced Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase 1 Part A: Dose escalation in patients with EGFR sensitizing mutation (Experimental): All eligible patients will receive the study treatment at selected oral dose(s) once daily, as per the assigned dose level from the pre-defined escalation scheme and SRC(Safety Review Committee) decision.
  Interventions: Drug: TRX-221
- Phase 1 Part B: 2 dose levels of TRX-221 in patients with EGFR sensitizing mutation (Experimental): All eligible patients will receive the study treatment at selected oral dose(s) once daily. Dose-levels will be selected from the Part A.
  Interventions: Drug: TRX-221
- Phase 2: Recommended Phase 2 dose(s) of TRX-221 in patients with EGFR C797X mutation (Experimental): All eligible patients will receive the study treatment at selected oral dose(s) once daily.
  Interventions: Drug: TRX-221

INTERVENTIONS:
Drug: TRX-221 — TRX-221 oral dose as defined

SUMMARY:
This is a Phase 1/2, open-label study designed to investigate the safety, tolerability, PK, and anti-tumor activity of the study treatment in the treatment of patients with EGFR mutant NSCLC, who progressed following prior standard treatments which include the approved EGFR-TKIs with activity against T790M (e.g., osimertinib).

DETAILED DESCRIPTION:
All eligible patients will receive the study treatment at selected oral dose(s) once daily. Patients will be treated continuously until disease progression or any other pre-defined discontinuation criteria are met.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with ECOG performance status score of 0 or 1
2. Histologically or cytologically confirmed diagnosis of relapsed or refractory, locally unresectable advanced or metastatic NSCLC harboring an activating EGFR mutation
3. Failed standard of care treatments progressed after anti tumor treatments including at least 1 approved EGFR TKI [Phase2: TKIs should include the approved EGFR TKIs with activity against T790M (e.g., osimertinib)]
4. Slots may be reserved for patients with certain resistant mutations (i.e., EGFR C797X mutation with or without T790M mutation as required by the sponsor) [Phase 1]
5. EGFR C797X mutation with or without T790M mutation [Phase 2]
6. Not received more than 1 prior line of platinum based chemotherapy in the metastatic setting [Phase 2]
7. Having at least 1 measurable tumor lesion per RECIST v1.1 criteria [Phase 2]
8. Having adequate bone marrow, hepatic, and renal function as specified in the protocol

Exclusion Criteria:

1. NSCLC with mixed cell histology or a tumor with histologic transformation of small cell elements
2. Patients having tumor with any additional known driver of alterations
3. Patients with presence of another active primary malignant tumor that has been diagnosed or required therapy within 2 years prior to the initiation of the study treatment
4. Patients who have unstable and symptomatic primary CNS tumors/metastasis, leptomeningeal metastases or spinal cord compression which are not suitable for enrollment, as judged by the Investigator
5. Patients having clinically active ongoing ILD of any etiology
6. Clinically significant cardiac conditions, infections, refractory GI diseases as specified in the protocol
7. Patients having any unresolved toxicities from prior anti tumor therapy and surgery greater than CTCAE Grade 1 at the time of starting the study treatment
8. Recent anticancer therapy: EGFR-TKI, Immunotherapy or any other systemic anticancer therapy or radiotherapy (specific duration prior to starting study medication per protocol)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Estimated)
Dates: Start 2024-06-14 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
[Phase1 PartA: Dose Escalation] To assess the safety/tolerability and determine the MTD/RP2D range of TRX-221 | Approx. 12 months
  Incidence and severity of AEs graded according to the NCI-CTCAE v5.0 Number and percentage of patients with TEAEs, SAEs, and DLTs Safety and tolerability as noted by laboratory data, vital signs, physical examinations, and 12-lead ECGs
[Phase1 PartB: Dose Exploration] To determine the RP2D of TRX-221 | Approx. 6-12 months
  Incidence and severity of AEs, TEAEs, SAEs Safety and tolerability as noted by laboratory data, vital signs, physical examinations, and 12-lead ECGs
[Phase2] To assess the anti-tumor activity of TRX-221 in patients with the selected EGFR-resistant mutation type | Approx. 6-12 months
  Tumor response rate (ORR)

SECONDARY OUTCOMES:
To characterize the PK profile of the study treatment | Throughout the study period, an average of 1 year
  Peak Plasma Concentration (Cmax)
To evaluate the preliminary anti-tumor activity of the study treatment (Phase 1) | Approx. 12 months
  ORR
To evaluate additional anti-tumor activity of the study treatment other than the primary endpoint (Phase 2) | Approx. 12 months
  PFS
To assess the safety and tolerability of the study treatment (Phase 2) | Approx. 12 months
  Incidence and severity of AEs, TEAEs, SAEs Safety and tolerability as noted by laboratory data, vital signs, physical examinations, and 12-lead ECGs

CONTACTS AND LOCATIONS:
Overall Officials: Therapex Co., Ltd Clinical Development, Study Director — Therapex Co., Ltd: Clinical Development
Locations (6):
- South Korea (6):
  - Seoul National University Bundang Hospital, Seongnam, Kyeongki
  - The Catholic University of Korea St. Vincent Hospital, Suwon, Kyeongki
  - Chungbuk National University Hospital, Chungju, North Chungcheong
  - Severance Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: No